CLINICAL TRIAL: NCT05926050
Title: The Acute Effects of a Dietary Supplement on Cognitive Performance in a Group of Highly Trained Athletes.
Brief Title: The Acute Effects of a Dietary Supplement on Cognitive Performance in Highly Trained Athletes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USANA Health Sciences (Industry)
Collaborators: U.S. Ski & Snowboard (Unknown)
Responsible Party: Principal Investigator, Mark Levy, Director of Product Validation, USANA Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202101CT
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Reaction Time
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled randomized clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement intervention (Experimental): Participants were treated with 2 tablets containing extracts of American ginseng, bacopa monnieri and coffee fruit
  Interventions: Dietary Supplement: Treatment (CopaPrime+ (USANA Health Sciences)
- Placebo Treatment (Placebo Comparator): Participants received 2 placebo tablets containing microcrystalline cellulose. The size, shape and appearance of the placebo tablet is identical to the treatment tablet.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Treatment (CopaPrime+ (USANA Health Sciences) — Participants received and consumed 2 treatment tablets immediately following baseline testing, and one hour prior to post-treatment testing. Each tablet contained extracts of Bacopa monnieri (150 mg), Coffea arabica (50 mg), and Panax quinquefolius L. (50 mg)
  Other Names: CopaPrime+ (USANA Health Sciences)
  Arms: Dietary supplement intervention
Other: Placebo — Participants received and consumed 2 placebo tablets immediately following baseline testing, and one hour prior to post-treatment testing. Each tablet contained microcrystalline cellulose. The size, shape and appearance of the placebo tablet was identical to the treatment tablet.
  Arms: Placebo Treatment

SUMMARY:
This study was designed to determine if a dietary supplement containing extracts of American ginseng, bacopa monnieri and coffee fruit can enhance cognitive performance in a population of trained athletes.

DETAILED DESCRIPTION:
In this study, we hypothesized that consumption of a dietary supplement containing extracts of American ginseng, bacopa monnieri and coffee fruit will improve reaction time and short-term memory in a population of highly trained athletes.

In order to test this hypothesis, we will employ a randomized, double blind, placebo controlled, parallel arm study design. 40-50 subjects will be recruited and randomized in a 1:1 ratio to either of two interventions:

Placebo: consumption of the placebo tablet Treatment: consumption of the supplement (treatment) tablet

On the day of the study, subjects will perform a series of reaction time tasks specific to the upper (i.e., arms) and lower (i.e., legs) body. They will also be asked to perform the stroop test. At the conclusion of baseline testing, subjects will consume either the placebo or treatment tablet. One hour later, the subjects will repeat all reaction time tasks as well as the stroop test. Differences in reaction time, as well as the error rate within each reaction time or stroop test, will serve as the primary endpoint. The data will then be analyzed to determine if there is a difference in the before and after reaction times and error rates between subjects on treatment and those consuming the placebo tablets.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed Informed Consent prior to screening for entry in the study
* Male or females between the ages of 18 and 30 (inclusive) without regard to race or ethnic background
* Are in generally good health and have no medical conditions that would prevent or interfere with their participation in the study
* Comprehensive Metabolic Panel results reported within normal laboratory reference ranges
* Have a Body Mass Index of ≤ 30
* Are fully able and willing to comply with the requirements of the study
* Are fully able and willing to keep scheduled appointments

Exclusion Criteria:

* Pregnant or attempting to become pregnant or lactating females.
* Chronic or acute use of prescription or over-the-counter medications that may interfere with absorption of the test supplement or confound results.
* Gastrointestinal conditions (e.g., inflammatory bowel disease, Crohn's disease, etc.) that may affect consumption of the treatment supplements.
* Significant acute or chronic illness or other medical conditions that will prevent or interfere with giving an informed consent, or with participation in the study; insulin-dependent and orally controlled diabetics will also be excluded from the study.
* Scheduling difficulties or lack of transportation that will prevent or interfere with their ability to attend all the necessary study visits.
* Individual's that have trouble swallowing pills.
* Individuals that have participated as a subject in any other clinical study within 30 days of the screening visit.
* A history of alcohol abuse or other substance abuse within the previous 2 years.
* Currently using tobacco products including chewing tobacco and cigarettes.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Reaction time | One hour
  Participants will perform a series of reaction time tasks prior to and after consumption of either the treatment or placebo tablets. Reaction times will be quantified and analyzed to determine if the intervention affected these measures.

SECONDARY OUTCOMES:
Stroop test | One hour
  Participants are asked to identify the font color of a word (i.e., red, blue, green, yellow) by pressing a specific key on the keyboard when the word appears on a computer screen. In situation #1, the font color of the word matches the written word (congruent test). In situation #2, the font color does not match the written word (incongruent test).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Levy, PhD, Principal Investigator — USANA Health Sciences
Locations (1):
- US Ski and Snowboard Center of Excellence, Park City, Utah, United States